CLINICAL TRIAL: NCT02630966
Title: A Randomized Double-Blind Phase 4 Study to Evaluate the Safety and Proportion of Subjects With Fistula Healing in 2 Dose Regimens of Entyvio (Vedolizumab IV) in the Treatment of Fistulizing Crohn's Disease (ENTERPRISE)
Brief Title: Vedolizumab IV 300 mg in the Treatment of Fistulizing Crohn's Disease
Acronym: ENTERPRISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vedolizumab-4003; 2015-000852-12 (EudraCT Number); U1111-1174-2252 (Registry Identifier: WHO)
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Crohn's Disease
Keywords: Drug therapy; Fistulizing Crohn´s disease; Perianal Fistula
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Vedolizumab IV 300 mg + Placebo (Experimental): Vedolizumab 300 mg, IV infusion, once, at Weeks 0, 2, 6, 14, and 22, and vedolizumab placebo-matching, IV infusion once, at Week 10 to maintain the blind.
  Interventions: Drug: Vedolizumab; Drug: Placebo
- Group 2: Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, IV infusion, once, at Weeks 0, 2, 6, 10, 14, and 22.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab 300 mg IV infusion
  Other Names: Entyvio; MLN0002; Kynteles
Drug: Placebo — 0.9% sodium chloride IV infusion
  Arms: Group 1: Vedolizumab IV 300 mg + Placebo

SUMMARY:
The purpose of this study is to evaluate the percentage of participants with perianal fistula healing at Week 30 in 2 different dose regimens of vedolizumab intravenous (IV) 300 milligram (mg) in participants with fistulizing Crohn's disease (CD).

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab IV. Vedolizumab IV is being tested to treat people who have fistulizing CD. This study will look at fistula healing in people who take vedolizumab IV.

The study is planned to enroll approximately 100 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Group 1: Vedolizumab IV 300 mg dose at Weeks 0, 2, 6, 14 and 22, and a placebo infusion at Week 10 (dummy inactive infusion - this is a solution that looks like the study drug but has no active ingredient).
* Group 2: Vedolizumab IV 300 mg dose at Weeks 0, 2, 6, 10, 14 and 22.

This multi-center trial will be conducted worldwide. The overall time to participate in this study from screening to 18 weeks after the last dose is 44 weeks. Participants will make multiple visits to the clinic, and will be contacted by telephone 6 months after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative has signed and dated a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has a diagnosis of CD established at least 3 months prior to randomization by clinical and endoscopic evidence and corroborated by a histopathology report.
4. Has a diagnosis of a minimum of 1 perianal draining fistula of at least 2 weeks duration as a complication of moderately to severely active CD, as identified on magnetic resonance image (MRI) at Screening. Other types of fistulae (enterocutaneous, abdominal) except rectovaginal fistulae are permitted, but the number of perianal draining fistulae is limited to 3.
5. All countries except France: The participant, historically, had an inadequate response with, lost response to, or was intolerant to either conventional therapy or a tumor necrosis factor-alpha (TNF-α) antagonist for their underlying CD (does not require treatment failure for currently active draining fistula).

   France only: The participant, historically, failed (ie, had an inadequate response with, lost response to, or was intolerant to) infliximab for treatment of their underlying CD or fistulizing CD.
6. If the participant had noncutting perianal seton placement as part of standard care, seton must be removed by Week 14 of the study.

Exclusion Criteria:

1. Has a diagnosis of ulcerative colitis or indeterminate colitis.
2. Has a perianal abscess greater than (>) 2 centimeter (cm) or an abscess that the investigator feels requires drainage based on either clinical assessment or MRI.
3. Has a Crohn's Disease Activity Index (CDAI) score >400.
4. Has an ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine.
5. Has significant anal or rectal stenosis.
6. Has active or latent tuberculosis (TB), regardless of treatment history.
7. Has evidence of active Clostridium difficile (C. difficile) infection or is having treatment for C. difficile infection or other intestinal pathogens during Screening.
8. Has current rectovaginal fistula.
9. Currently has more than 3 draining perianal fistulae. Note: Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (18):
- United States (3):
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - GIRI (GI Research Institute), Vancouver, British Columbia
- France (4):
  - CHRU de Lille - Hopital Claude Huriez, Lille
  - Hopital l'Archet II, Nice
  - CHU de Rennes - Hopital de Pontchaillou, Rennes
  - Hopital de Brabois, Vandœuvre-lès-Nancy
- Italy (2):
  - Azienda Ospedaliera S. Orsola-Malpighi, Bologna
  - Istituto Clinico Humanitas IRCCS, Milan
- Netherlands (3):
  - Academic Medical Center, Amsterdam
  - Leids Universitair Medisch Centrum, Leiden
  - Erasmus MC, Rotterdam
- Spain (2):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario y Politecnico La Fe, Valencia
- United Kingdom (2):
  - Nottingham University Hospitals NHS Trust, Nottingham
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Schwartz DA, Peyrin-Biroulet L, Lasch K, Adsul S, Danese S. Efficacy and Safety of 2 Vedolizumab Intravenous Regimens for Perianal Fistulizing Crohn's Disease: ENTERPRISE Study. Clin Gastroenterol Hepatol. 2022 May;20(5):1059-1067.e9. doi: 10.1016/j.cgh.2021.09.028. Epub 2021 Sep 29. PMID 34597729

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 13 investigative sites in Canada, France, Italy, the Netherlands, Spain, the United Kingdom, and the United States from 10 August 2016 to 14 November 2018.
Pre-assignment Details: Participants with diagnosis of moderately to severely active Crohn's disease and 1 to 3 draining perianal fistula(e) of at least 2 weeks duration were randomized in 1:1 ratio to receive vedolizumab IV 300 mg dose at Weeks 0,2,6,14,22 and vedolizumab placebo-matching IV dose at Week 10 or vedolizumab IV 300 mg dose at Weeks 0,2,6,10,14,and 22.
Period: Overall Study
Arm/Group | Group 1: Vedolizumab IV 300 mg + Placebo | Group 2: Vedolizumab 300 mg
Started | 16 | 18
Completed (Completed here refers to participants who completed study drug.) | 14 | 10
Not Completed | 2 | 8
Not completed — Adverse Event | 1 | 3
Not completed — Significant Protocol Deviation | 0 | 2
Not completed — Voluntary Withdrawal | 1 | 1
Not completed — Lack of Efficacy | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Vedolizumab IV 300 mg + Placebo | Group 2: Vedolizumab 300 mg | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (10.35) | 35.1 (10.67) | 35.1 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 14 | 15 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 15 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1 | 0 | 1
  France | 2 | 3 | 5
  Italy | 5 | 6 | 11
  Netherlands | 2 | 3 | 5
  Spain | 3 | 2 | 5
  United Kingdom | 1 | 1 | 2
  United States | 2 | 3 | 5
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 170.1 (6.35) | 176.4 (10.38) | 173.4 (9.17)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 73.65 (15.986) | 68.36 (14.661) | 70.85 (15.299)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg per square meter (kg/m^2)] — Body Mass Index=weight/[height^2]
  kg per square meter (kg/m^2) | 25.40 (5.080) | 21.84 (3.580) | 23.52 (4.646)
Smoking Classification [Count of Participants; unit: Participants]
  Never-smoker | 7 | 8 | 15
  Current smoker | 7 | 4 | 11
  Ex-smoker | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 50% Reduction From Baseline in the Number of Draining Perianal Fistulae (of Those Draining at Baseline)
Description: Closed fistulae are no longer draining despite gentle finger compression.
Time Frame: Baseline, Week 30
Population: Modified Full Analysis Set (mFAS) included all participants in FAS who had at least one draining fistula at baseline (Day 1). FAS included all randomized participants who received at least 1 dose of study medication and have a post baseline assessment of fistula healing. Data is reported for participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Vedolizumab IV 300 mg + Placebo | Group 2: Vedolizumab 300 mg
Number analyzed (Participants) | 12 | 8
percentage of participants | 75.0 [50.5 to 99.5] | 75.0 [45.0 to 100.0]

2. Secondary Outcome: Percentage of Participants With at Least 50% Reduction of From Baseline in the Number of Draining Perianal Fistulae (of Those Draining at Baseline) at Both Weeks 22 and 30
Description: Closed fistulae are no longer draining despite gentle finger compression.
Time Frame: Weeks 22 and 30
Population: The mFAS includes all participants in the FAS who had at least one draining fistula at baseline (Day 1). The FAS includes all randomized participants who received at least 1 dose of study medication and have a post baseline assessment of fistula healing. Data is reported for participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Vedolizumab IV 300 mg + Placebo | Group 2: Vedolizumab 300 mg
Number analyzed (Participants) | 11 | 8
percentage of participants | 72.7 [46.4 to 99.0] | 62.5 [24.5 to 91.5]

3. Secondary Outcome: Percentage of Participants With 100% Perianal Fistulae Closure (of the Fistulae Draining at Baseline)
Description: Closed fistulae are no longer draining despite gentle finger compression.
Time Frame: Week 30
Population: The mFAS included all participants in the FAS who had at least one draining fistula at baseline (Day 1). The FAS included all randomized participants who received at least 1 dose of study medication and have a post baseline assessment of fistula healing. Data is reported for participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Vedolizumab IV 300 mg + Placebo | Group 2: Vedolizumab 300 mg
Number analyzed (Participants) | 12 | 8
percentage of participants | 58.3 [30.4 to 86.2] | 62.5 [24.5 to 91.5]

4. Secondary Outcome: Time to First Perianal Fistulae Closure (of Those Fistulae Draining at Baseline)
Description: Closed fistulae are no longer draining despite gentle finger compression.The time to first fistula closure was analyzed descriptively using Kaplan-Meier product limit methods, with participants for which no fistula closure is reported being censored at the time of their last fistulae assessment or date of last record (Week 30 or early discontinuation). Estimated median time to fistula closure (and 95%CI) are reported.
Time Frame: Up to Week 30
Population: mFAS included participants in FAS with >=1 draining fistula at baseline (Day 1). FAS included all randomized participants who received >=1 dose of study drug, have a post baseline assessment of fistula healing.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Group 1: Vedolizumab IV 300 mg + Placebo | Group 2: Vedolizumab 300 mg
Number analyzed (Participants) | 14 | 14
days | 30.5 [15.0 to 71.0] | 159.0 [16.0 to NA] — Upper limit of 95% of confidence interval (CI) was not estimable due to low number of participants with events.

5. Secondary Outcome: Time to Last (100%) Perianal Fistulae Closure (of Those Fistulae Draining at Baseline)
Description: Closed fistulae are no longer draining despite gentle finger compression. The time to first fistula closure was analyzed descriptively using Kaplan-Meier product limit methods, with participants for which no fistula closure is reported being censored at the time of their last fistulae assessment or date of last record (Week 30 or early discontinuation). Estimated median time to fistula closure (and 95%CI) are reported.
Time Frame: Up to Week 30
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Group 1: Vedolizumab IV 300 mg + Placebo | Group 2: Vedolizumab 300 mg
Number analyzed (Participants) | 14 | 14
days | 45.0 [15.0 to 155.0] | 159.0 [16.0 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events.

6. Secondary Outcome: Duration of Perianal Fistulae Response (of Those Fistulae Draining at Baseline)
Description: Duration of fistula response was measured by number of days with/without drainage. Duration of perianal fistula response (days) was derived as the sum of days with perianal fistula response between Day 1 and the end of the study (Week 30 or early discontinuation). Perianal fistula response is defined as reduction in the number of draining perianal fistulae (of those draining at Baseline) draining of at least 50%.
Time Frame: Up to Week 30
Population: The mFAS included all participants in the FAS who had at least one draining fistula at baseline (Day 1). The FAS included all randomized participants who received at least 1 dose of study medication and have a post baseline assessment of fistula healing.
Measure: Median (Full Range); unit: days
Arm/Group | Group 1: Vedolizumab IV 300 mg + Placebo | Group 2: Vedolizumab 300 mg
Number analyzed (Participants) | 14 | 14
days | 158.5 [0 to 202] | 33.5 [0 to 203]

ADVERSE EVENTS:
Time Frame: Up to approximately 44 weeks
Description: At each visit investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by investigator was recorded, irrespective of relation to study treatment. Safety Analysis Set included all participants who received at least 1 dose of study medication.
Arm/Group | Group 1: Vedolizumab IV 300 mg + Placebo | Group 2: Vedolizumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 4/16 | 3/18
Other Adverse Events (participants affected / at risk) | 15/16 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Vedolizumab IV 300 mg + Placebo (N=16) | Group 2: Vedolizumab 300 mg (N=18)
Crohn's disease (Gastrointestinal disorders) | 1 | 1
Ileal stenosis (Gastrointestinal disorders) | 1 | 0
Hyperpyrexia (General disorders) | 0 | 1
Anal abscess (Infections and infestations) | 3 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Vedolizumab IV 300 mg + Placebo (N=16) | Group 2: Vedolizumab 300 mg (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 2 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0
Rectal discharge (Gastrointestinal disorders) | 0 | 1
Rectal stenosis (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 5
Toothache (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Abdominal tenderness (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Dyschezia (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 2 | 2
Subileus (Gastrointestinal disorders) | 0 | 1
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Oral pain (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 4
Influenza like illness (General disorders) | 1 | 0
Catheter site bruise (General disorders) | 1 | 0
Granuloma (General disorders) | 1 | 0
Anal abscess (Infections and infestations) | 3 | 0
Anal fistula infection (Infections and infestations) | 0 | 1
Campylobacter infection (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Perineal abscess (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Rhinitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 4
Migraine (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Device expulsion (Product Issues) | 0 | 1
Device loosening (Product Issues) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Skin striae (Skin and subcutaneous tissue disorders) | 1 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Takeda decided to close enrollment after randomizing 34 participants.Decision was taken due to challenges in recruitment and was not related to any safety concerns.Participants randomized before enrollment closure continued participation as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT02630966/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT02630966/SAP_001.pdf